CLINICAL TRIAL: NCT04181671
Title: Effects of Low Resistance Venous Blood Flow Restriction Training (LR-VBFRT) on Biceps Brachii Muscle Performance
Brief Title: Low Resistance Venous Blood Flow Restriction Training (LR-VBFRT) on Biceps Brachii Muscle Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU 00563
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Muscle Weakness Condition
Keywords: Exercise Training

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated at the same time following their respective protocols
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Resistance Training Group (Experimental): The experimental group will receive low resistance blood flow restriction training with 30% of 1 RM.
  Interventions: Other: Low Resistance training with venous blood flow restriction
- High Resistance Training Group (Active Comparator): Participants of this group will receive High resistance training (80% of 1 RM) without blood flow restriction.
  Interventions: Other: High Resistance training

INTERVENTIONS:
Other: Low Resistance training with venous blood flow restriction — Total 20 males will participate in this group after warmup , Blood flow restriction will be provided through sphygmomanometer optimum pressure will be measured through following formula occlusion pressure (mmHg) = 0.514 (SBP) + 0.339 (DBP) + 1.461 (Arm circumference) + 17.236 then 30% of 1RM will be used for training . The standard protocol will be used which is four sets (1st set-30 repetitions, 2nd set-15 repetitions, 3rd set-15 repetitions, and 4th set-15 repetitions) with 30-60 s of interval between sets. ( the cuff must be deflated between sets of exercise) for 8 weeks (24) sessions on non-consecutive days. participants will be re-assessed for all baseline variables after 8 weeks of training biceps curls will be used for training.
  Heart Rate and oxygen saturation will be measured during the session through Pulse oximeter
  Arms: Low Resistance Training Group
Other: High Resistance training — Total 20 males will participate in this group after warm up. 80% of 1RM will be used for training, 3 sets of 8 repetitions will be used with 30-60 s of interval between sets. for 8 weeks (24) sessions on non-consecutive days.No blood flow restriction will be applied to this group Participants will be re-assessed for all baseline variables after 8 weeks of training. Bicep curls will be used for training.
  Arms: High Resistance Training Group

SUMMARY:
Resistance training has been widely recognized as an effective stimulus for increasing skeletal muscle size and strength. This study intends to compare the effects of high resistance training without blood flow restriction and the low resistance training with blood flow restriction training on bicep muscle performance.

DETAILED DESCRIPTION:
The study is Randomized Control Trail, which is being conducted in RIPHAH COLLEGE OF REHABILITATION SCIENCES. Sample size of 40 individual was calculated using Epitool with 95% confidence interval (CI) and power 80%. Individual will be screened out according to inclusion criteria. Individuals will be allocated randomly into two groups, 20 in high resistance training group and 20 in low resistance training with blood flow restriction group by sealed envelope method.

High resistance training will be use in control group.Low resistance with blood flow restriction training will be used in experimental group.

Assessment will be done on baseline 2-4 days prior to the intervention and after 8 weeks of training.

Data will be analyzed on SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age: 20-28 year
* Body mass index: 18.5-24.9

Exclusion Criteria:

* Vascular Disease
* Upper Limb Pathology Requiring Surgical Intervention
* Upper Limb Musculoskeletal Issues
* Blood Pressure >140/90
* Coronary Artery Disease
* Venous Thromboembolism
* Congenital Cardiac Diseases
* Syncope, Arrhythmias, Smokers
* Alcohol Use
* Supplements Intake
* whey Protein Intake

Ages: 20 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants are recruited in the study.
Enrollment: 40 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Baseline
  Handheld dynamometer will be used for measuring muscle strength of bicep muscle of all participants by single examiner
Muscle strength | Post 6 weeks
  Handheld dynamometer will be used for measuring muscle strength of bicep muscle of all participants by single examiner
1 Repetition maximum | Baseline
  1RM will be assess using Epley's formula of 1RM , RM= w(1+r/30) where "w" is the sub maximal weight and "r" is repetition then percentages of 1RM will be used for training purposes 80% of 1 RM for control group and 30% of 1RM for experimental group.
1 Repetition maximum | Post 6 weeks
  1RM will be assess using Epley's formula of 1RM , RM= w(1+r/30) where "w" is the sub maximal weight and "r" is repetition then percentages of 1RM will be used for training purposes 80% of 1 RM for control group and 30% of 1RM for experimental group.
Bicep Muscle power | Baseline
  Muscle power will be assesses of all the participants using power formula(Power= W/t= FS/t) for that force (F) will be assessed through dynamometer in newton covered distance (S) will be taken as covered range of motion and will be asses through goniometer (elbow flexion in supinated position). Time (t) will be calculated using stop watch
Bicep Muscle power | Post 6 weeks
  Muscle power will be assesses of all the participants using power formula(Power= W/t= FS/t) for that force (F) will be assessed through dynamometer in newton covered distance (S) will be taken as covered range of motion and will be asses through goniometer (elbow flexion in supinated position). Time (t) will be calculated using stop watch
Bicep muscle endurance testing | Baseline
  Bicep muscle endurance will be calculated prior to the intervention by asking participants to lift light -moderate weight and perform bicep curls in supinated position the total number of repetition they will perform doing complete eccentric and concentric movement of the muscle will be taken as the endurance of the bicep muscle
Bicep muscle endurance testing | Post 6 weeks
  Bicep muscle endurance will be calculated prior to the intervention by asking participants to lift light -moderate weight and perform bicep curls in supinated position the total number of repetition they will perform doing complete eccentric and concentric movement of the muscle will be taken as the endurance of the bicep muscle
Arm circumference | Baseline
  arm circumference will be measured in centimeters at the midpoint between the acromion process and the center of the elbow(by measuring tape)
Arm circumference | Post 6 weeks
  arm circumference will be measured in centimeters at the midpoint between the acromion process and the center of the elbow(by measuring tape)

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- RCRAHS Potohar campus, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos GE, Luecke TJ, Wendeln HK, Toma K, Hagerman FC, Murray TF, Ragg KE, Ratamess NA, Kraemer WJ, Staron RS. Muscular adaptations in response to three different resistance-training regimens: specificity of repetition maximum training zones. Eur J Appl Physiol. 2002 Nov;88(1-2):50-60. doi: 10.1007/s00421-002-0681-6. Epub 2002 Aug 15. PMID 12436270
- [Background] Lixandrao ME, Ugrinowitsch C, Laurentino G, Libardi CA, Aihara AY, Cardoso FN, Tricoli V, Roschel H. Effects of exercise intensity and occlusion pressure after 12 weeks of resistance training with blood-flow restriction. Eur J Appl Physiol. 2015 Dec;115(12):2471-80. doi: 10.1007/s00421-015-3253-2. Epub 2015 Sep 1. PMID 26323350
- [Background] Mattar MA, Gualano B, Perandini LA, Shinjo SK, Lima FR, Sa-Pinto AL, Roschel H. Safety and possible effects of low-intensity resistance training associated with partial blood flow restriction in polymyositis and dermatomyositis. Arthritis Res Ther. 2014 Oct 25;16(5):473. doi: 10.1186/s13075-014-0473-5. PMID 25344395
- [Background] Wilson JM, Lowery RP, Joy JM, Loenneke JP, Naimo MA. Practical blood flow restriction training increases acute determinants of hypertrophy without increasing indices of muscle damage. J Strength Cond Res. 2013 Nov;27(11):3068-75. doi: 10.1519/JSC.0b013e31828a1ffa. PMID 23446173
- [Background] Loenneke JP, Allen KM, Mouser JG, Thiebaud RS, Kim D, Abe T, Bemben MG. Blood flow restriction in the upper and lower limbs is predicted by limb circumference and systolic blood pressure. Eur J Appl Physiol. 2015 Feb;115(2):397-405. doi: 10.1007/s00421-014-3030-7. Epub 2014 Oct 22. PMID 25338316